CLINICAL TRIAL: NCT06579404
Title: An Open-label, Multinational, Multicentre, Randomised, Single-period Parallel Study to Assess the Efficacy, Safety and Utility of Fully Closed-loop Insulin Delivery Compared to Standard Insulin Therapy With CGM in Adults With Type 2 Diabetes
Brief Title: Closed-loop in Adults With Type 2 Diabetes
Acronym: COYOTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: University of Edinburgh (Other); Jaeb Center for Health Research (Other); Swansea University (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Professor of Metabolic Technology, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COYOTE
Record Dates: First submitted 2024-08-16; First posted 2024-08-30 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Closed-loop insulin delivery; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A multicentre, multinational, open-label, randomised single period, parallel design study contrasting fully closed-loop insulin delivery and standard insulin therapy with CGM over 26 weeks in adults with type 2 diabetes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fully closed-loop insulin delivery (CamAPS HX) (Experimental): The automated closed loop system (CamAPS FX) will consist of:
  * YpsoPump insulin pump (Ypsomed, Burgdorf, Switzerland)
  * FreeStyle Libre 3 glucose sensor (Abbott Diabetes Care, CA, USA)
  * Smartphone hosting CamAPS HX app with the Cambridge model predictive control algorithm
  * Cloud upload system to review CGM/insulin data.
  Participants will use the fully closed-loop system for 26 weeks at home
  Interventions: Device: CamAPS HX
- Standard insulin therapy with glucose sensor (Active Comparator): Usual insulin therapy and FreeStyle Libre 3 glucose sensor (Abbott Diabetes Care, CA, USA) for 26 weeks at home.
  Interventions: Other: Standard insulin therapy with glucose sensor

INTERVENTIONS:
Device: CamAPS HX — The automated closed loop system (CamAPS HX) will consist of:
  YpsoPump insulin pump Freestyle Libre 3 glucose sensor Smartphone hosting CamAPS HX app with the Cambridge model predictive control algorithm
  Arms: Fully closed-loop insulin delivery (CamAPS HX)
Other: Standard insulin therapy with glucose sensor — Participants usual insulin therapy with Freestyle Libre 3 glucose sensor
  Arms: Standard insulin therapy with glucose sensor

SUMMARY:
The main objective of this study is to determine the efficacy, safety and utility of fully closed-loop glucose control in the home setting in adults with type 2 diabetes (T2D). This study builds on previous and on-going studies of closed-loop systems that have been performed in Cambridge in adults with type 2 diabetes in the inpatient and in the home setting and in children and adults with type 1 diabetes.

This is an open-label, multi-national, multi-centre, randomised, single-period parallel study, involving a run-in period followed by a 26-week intervention period during which glucose levels will be controlled either by a fully closed-loop system or by participants usual insulin therapy with continuous glucose monitoring. A total of up to 224 adults with type 2 diabetes using insulin will be recruited through outpatient diabetes clinics, primary care centres, social media advertising and other established methods at participating centres. Participants will receive appropriate training in the safe use of the study devices.

The primary outcome is the between group difference in HbA1c at 26 weeks. Other key outcomes include the time spent with glucose levels within, above and below the target glucose range (3.9-10.0mmol/L) and mean sensor glucose as recorded by CGM over the 26 weeks. Insulin requirements, body weight, renal and liver function will also be compared. Safety evaluation comprises severe hypoglycaemic episodes, and other adverse and serious adverse events. Human factors outcomes include CGM & closed-loop usage, questionnaires and semi-structured interviews.

DETAILED DESCRIPTION:
Purpose of clinical trial:

To determine the efficacy, safety and utility of fully closed-loop insulin delivery over 26 weeks in the home setting in adults with type 2 diabetes.

Study objectives:

To determine the efficacy, safety and utility of fully closed-loop insulin delivery over 26 weeks in the home setting in adults with type 2 diabetes.

1. EFFICACY: The objective is to assess the ability of fully closed-loop insulin delivery to improve glucose control as measured by HbA1c (primary endpoint) and sensor glucose metrics.
2. SAFETY: The objective is to evaluate the safety of fully closed-loop insulin delivery in terms of episodes and severity of hypoglycaemia, and nature and severity of other adverse events.
3. UTILITY: The objective is to determine the acceptability and duration of use of the CGM and closed-loop system.
4. HUMAN FACTORS: The objective is to assess cognitive, emotional, and behavioural characteristics of participants and their response to the closed-loop system using validated questionnaires and semi-structured interviews.

   Participating clinical centres:

   UK - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust. - Imperial College Healthcare NHS Trust, London

   - Manchester Royal Infirmary, Manchester University NHS Foundation Trust

   - King's College Hospital, King's College Hospital NHS Foundation Trust, London

   - Guy's and St Thomas' NHS Foundation Trust

   - Norfolk and Norwich University Hospital, Norfolk and Norwich University Hospitals NHS Foundation Trust

   - University Hospitals of Leicester NHS Trust

   Switzerland

   - Inselspital, Bern University Hospital, Bern

   France

   - Centre Hospitalier Universitaire (CHU) de Toulouse

   Germany

   - Medical Center - University of Freiburg

   Austria

   - Medical University of Graz, Graz

   Czech Republic

   - Diabetes Centre, Institute for Clinical and Experimental Medicine, Prague

   Sample Size:

224 participants (112 per group) will be randomised. Recruitment will target a minimum quota of 25% of participants using basal insulin and a minimum quota of 60% of participants using multiple daily insulin injections.

Maximum duration of study for a subject: 30 weeks

Recruitment:

Participants will be recruited through outpatient diabetes clinics, primary care centres, social media advertising or other established methods at participating centres

Consent:

Participants will be asked to provide written informed consent.

Baseline Assessment:

Eligible participants will undergo baseline evaluation involving talking a medical history including demographics, height/weight, waist hip ratio and blood pressure measurement and blood samples for HbA1c, fasted lipid profile, renal and liver function. A urine albumin-creatinine ratio (ACR) will be performed, along with a urine pregnancy test in females of child-bearing age. Human factors questionnaires will be completed and a masked glucose sensor will be applied.

Run-in Period:

During a 2-3 week run-in period, participants will use their usual insulin therapy and wear a masked CGM system. At the end of the run-in period, for compliance, at least 10 days of CGM data needs to be recorded. CGM data during the run-in period will be used to assess baseline glucose control before the start of the intervention phase.

Randomisation:

Eligible participants will be randomised in a 1:1 ratio using central randomisation software to fully closed-loop or standard insulin therapy with CGM for 26 weeks. Randomisation will be stratified by site and baseline HbA1c.

Fully closed loop insulin delivery (intervention arm):

Following randomisation, participants in the closed-loop group will receive training on the study CGM, study insulin pump and closed-loop App during a 1-2 hour outpatient session. Competency on the use of the closed-loop system will be evaluated. Further training may be delivered as required. Participants will be advised to use the closed-loop system for the next 26 weeks.

Standard insulin therapy with CGM (control arm):

Following randomisation, participants in the control group will use their usual insulin therapy and the study CGM. Training on the use of the CGM will be provided. Participants will use standard insulin therapy and CGM for the next 26 weeks.

3 month study visit: Weight, waist hip ratio and blood pressure will be measured and a blood sample will be taken for measurement of HbA1c, fasted lipid profile, renal and liver function. Data from the closed-loop system and CGM system will be reviewed. Human factors questionnaires will be completed.

End of study assessments:

Weight, waist hip ratio and blood pressure will be measured and a blood sample will be taken for measurement of HbA1c, fasted lipid profile, renal and liver function. Urinary ACR will be measured. Human factors questionnaires will be completed and a subset of participants will participate in interviews. Study devices will be returned and participants will resume their usual insulin therapy and standard glucose monitoring.

Procedures for safety monitoring during trial:

Standard operating procedures for monitoring and reporting of all adverse events and adverse device events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

A data safety and monitoring board (DSMB) will be informed of all serious adverse events and any unanticipated serious adverse device effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of subjects on safety grounds:

A participant may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

* Participant is unable to demonstrate safe use of study devices as judged by the investigator
* Serious adverse events
* Significant protocol violation or non-compliance
* Decision by the investigator, or the Sponsor, that termination is in the participant's best medical interest
* Pregnancy, planned pregnancy, or breast feeding
* Allergic reaction to insulin or severe allergic reaction to adhesive surface of infusion set or glucose sensor
* Technical grounds (e.g. participant relocates)

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Type 2 diabetes diagnosed for at least 12 months
* Established on an SGLT2 inhibitor and/or GLP-1 receptor agonist for at least 3 months, or have been offered these therapies previously.
* Treatment with insulin therapy for at least 6 months
* HbA1c ≤ 15% (140 mmol/mol) analysis from local laboratory or equivalent
* Willing to wear study devices and follow study instructions
* Capacity to consent to participate in the study

Exclusion Criteria:

* Type 1 diabetes
* Current use of insulin pump
* Current use of any closed-loop system
* Any physical/psychological disease or medication(s) likely to interfere with the conduct of the study and interpretation of the study results, as judged by study clinician
* Known or suspected allergy against insulin
* Medically documented allergy towards the adhesive
* Pregnancy, planned pregnancy, or breast feeding
* Severe visual impairment
* Severe hearing impairment
* Medically documented allergy towards the adhesive (glue) of plasters
* Serious skin diseases located at places of the body, which potentially are possible to be used for localisation of the glucose sensor
* Illicit drugs abuse
* Prescription drugs abuse
* Alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) at 26 weeks | at 26 weeks
  Centralised measurement of HbA1c

SECONDARY OUTCOMES:
Proportion of time spent in target glucose range (3.9 to 10.0mmol/L) | over 26 weeks
  Sensor glucose metric measured as a %
Mean glucose (mmol/L) | over 26 weeks
  Sensor glucose metric measured in mmol/L
Proportion of time spent above target glucose (>10.0mmol/l) | over 26 weeks
  Sensor glucose metric measured as a %
Proportion of time spent below target glucose (<3.9mmol/L) | over 26 weeks
  Sensor glucose metric measured as a %
Standard deviation of sensor glucose | over 26 weeks
  Sensor glucose metric measured in mmol/L
Coefficient of variation of sensor glucose | over 26 weeks
  Sensor glucose metric measured as a %
Proportion of time spent below target glucose (<3.5mmol/L) | over 26 weeks
  Sensor glucose metric measured as a %
Proportion of time spent below target glucose (<3.0mmol/L) | over 26 weeks
  Sensor glucose metric measured as a %
Proportion of time spent above target glucose (>13.9mmol/l) | over 26 weeks
  Sensor glucose metric measured as a %
Proportion of time spent above target glucose (>16.7mmol/l) | over 26 weeks
  Sensor glucose metric measured as a %
Proportion of time spent above target glucose (>20.0mmol/l) | over 26 weeks
  Sensor glucose metric measured as a %
Proportion of participants with HbA1c <7.0% [53mmol/mol] (%) | at 26 weeks
  Binary metric of HbA1c
Proportion of participants with HbA1c <7.5% [58mmol/mol] (%) | at 26 weeks
  Binary metric of HbA1c
Total daily insulin dose | over 26 weeks
  Measured in units/day
Body weight | at 26 weeks
  Measured in kilograms
Waist hip ratio | 26 weeks
  Ratio
Body Mass Index (BMI) | 26 weeks
  Measured in kg/m2
Fasted lipid profile | 26 weeks
  Measured in mmol/L
Renal function | 26 weeks
  Renal function as measured by serum creatinine
Renal function | 26 weeks
  Renal function as measured by estimated Glomerular Filtration Rate
Renal function | 26 weeks
  Renal function as measured by urinary albumin creatinine ratio
Liver function | 26 weeks
  Liver function as measured by FIB4 index
Liver function | 26 weeks
  Liver function as measured by alanine transaminase (ALT)
Liver function | 26 weeks
  Liver function as measured by aspartate transaminase (AST)
Liver function | 26 weeks
  Liver function as measured by alkaline phosphatase (ALP)
Liver function | 26 weeks
  Liver function as measured by gamma-glutamyl transferase (yGT)
Liver function | 26 weeks
  Liver function as measured by serum bilirubin
Liver function | 26 weeks
  Liver function as measured by albumin and FIB4 index

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, Principal Investigator — University of Cambridge
Locations (12):
- University of Melbourne, Melbourne, Australia
- Medical University of Graz, Graz, Austria
- Diabetes Centre, Institute of Clinical and Experimental Medicine, Prague, Czechia
- CHU de Toulouse, Toulouse, France
- Bern University Hospital, Bern, Switzerland
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Derby Hospital, Derby
  - Leicester Diabetes Centre, Leicester
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital, King's College NHS Foundation Trust, London
  - Manchester Royal Infirmary, Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.